CLINICAL TRIAL: NCT03150771
Title: A Phase 1, Open-label, Single Ascending Dose, Parallel Arm Trial to Determine the Pharmacokinetics, Safety, and Tolerability of Aripiprazole 2 Month Intramuscular Depot Administered Gluteally in Adult Subjects With Schizophrenia
Brief Title: Study to Determine the Pharmacokinetics, Safety & Tolerability of Aripiprazole in Adults With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 031-201-00104
Record Dates: First submitted 2017-05-02; First posted 2017-05-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Aripiprazole; single; gluteal
  Interventions: Drug: Aripiprazole
- Cohort 2 (Experimental): Aripiprazole; single; gluteal
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Injection
  Other Names: Abilify Maintena

SUMMARY:
This trial will determine the Pharmacokinetics, safety and tolerability of single-dose Aripiprazole administered intramuscularly in adults with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Male and female individuals between 18 and 64 years, inclusive, at screening with a current diagnosis of schizophrenia as defined by Diagnostic and Statistical Manual of Mental Disorders: edition 5 (DSM-5)
* Body mass index (BMI) between 18 and 35 kg/m^2 at screening
* Male and female subjects who are surgically sterile, female subjects who have been postmenopausal for at least 12 consecutive months prior to screening or male/female subjects who agree to remain abstinent or practice 2 of the approved birth control methods from screening for at least 150 days after dose of Investigational Medical Product (IMP) for female subjects or 180 days after dose of IMP for male subjects.
* Documented history of previously tolerating Aripiprazole per investigator's judgment.

Exclusion Criteria:

* Met DSM-5 criteria for substance use disorder within past 180 days
* Positive drug screen for drugs of abuse
* Use of more than 1 antipsychotic medication at screening or baseline, except for oral Aripiprazole administered during tolerability testing and current antipsychotic medication
* Subjects may not receive varenicline beyond the screening visit.
* Subjects who had participated in any clinical trial involving a psychotropic medication within 1 month prior to administration of IMP
* Major surgery within 30 days prior to administration of IMP or surgery during the trial
* Subjects at significant risk of committing suicide based on history, psychiatric exams
* Subjects currently in an acute relapse of schizophrenia
* Subjects with a current DSM-5 diagnosis other than schizophrenia
* Subjects with a history of neuroleptic malignant syndrome, seizure disorder, or clinically significant tardive dyskinesia
* Subjects who have had electroconvulsive therapy within 2 months prior to administration of IMP
* Females who are breast-feeding and/or who have a positive pregnancy test result prior to receiving IMP
* History of or current hepatitis or Acquired Immunodeficiency Syndrome or carriers of Hepatitis B surface antigen (HBsAG), Hepatitis C antigen (anti-HCV) and/or Human Immunodeficiency Virus (HIV) antibodies

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) [safety and tolerability] | Screening Days -30 to Day 182 post dose/Early Termination
  AEs will be monitored to assess safety and tolerability of drug
Clinical Laboratory Tests [safety and tolerability] | Screening Days -30 to Day 182 post dose/Early Termination
  Hematology, clinical chemistry & urinalysis tests will be performed to assess the safety and tolerability of drug.
Electrocardiograms (ECGs) [Safety and tolerability] | Screening Days -30 to Day 182 post dose/Early Termination
  Heart rate, RR, PR, WRS and WT intervals will be monitored to assess the safety and tolerability of the drug.
Vital Signs [safety and tolerability] | Screening Days -30 to Day 182 post dose/Early Termination
  Systolic/diastolic blood pressure, heart rate and body temperature will be monitored to assess the safety and tolerability of the drug.
Suicidality via Columbia-Suicide Severity Rating Scale (C-SSRS) [safety and tolerability] | Screening Days -30 to Day 182 post dose/Early Termination
  C-SSRS score will be monitored throughout the trial to assess the safety and tolerability of drug
Extrapyramidal Symptoms (EPS) Rating Scales | Screening Days -30 to Day 182 post dose/Early Termination
  EPS score will be monitored to assess safety and tolerability of drug
Investigator's Assessment of Injection Site | Screening Days -30 to Day 182 post dose/Early Termination
  The injection site will be monitored to assess the safety and tolerability of drug
Visual Analog Scale (VAS) Scores for Pain Perception | Day 1 to Day 28 post dose
  VAS score will be monitored to assess safety and tolerability of drug

SECONDARY OUTCOMES:
Pharmacokinetics - Maximum plasma concentration (Cmax) | Day 1 to Day 182/Early Termination
  The maximum plasma concentration of drug at injection site will be assessed for plasma Aripiprazole and its major metabolite dehydro-aripiprazole
Pharmacokinetics - time of maximum plasma concentration (tmax) | Day 1 to Day 182/Early Termination
  The amount of time that the maximum plasma concentration of drug at injection site will be assessed for plasma Aripiprazole and its major metabolite dehydro-aripiprazole
Pharmacokinetics - area under concentration-time curve (AUC) calculated from time zero to time t (AUCt) | Day 1 to Day 182/Early Termination
  AUCt will be assessed for plasma Aripiprazole and its major metabolite dehydro-aripiprazole to determine average concentration of drug over time
Pharmacokinetics - AUC calculated from time to infinity | Day 1 to Day 182/Early Termination
  AUCinfinity will be assessed for plasma Aripiprazole and its major metabolite dehydro-aripiprazole to determine total drug exposure over time
Pharmacokinetics - Terminal-phase elimination half-life (t1/2,z) | Day 1 to Day 182/Early Termination
  t1/2,z will be assessed for plasma Aripiprazole and its major metabolite dehydro-aripiprazole to determine drug persistence in the body

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Woodland International Research Group, Little Rock, Arkansas
  - CNRI-San Diego, San Diego, California
  - Community Clinical Research Inc., Austin, Texas